CLINICAL TRIAL: NCT06900868
Title: The Effect of Bulk Filling Flowable Composite on Caries Recurrence in Deep Marginal Elevation: a Randomized Clinical Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Future University in Egypt (Other)
Responsible Party: Principal Investigator, AHMED AYMAN ESMAIL MAHMOUD, Principal investigator, Future University in Egypt
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Deep marginal elevation
Record Dates: First submitted 2025-03-22; First posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: DME; Dental Caries; Dental; Deep Margin Elevation
Keywords: Deep margin elevation
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- arm (Active Comparator): Beautifil-Bulk Flowable Deep margin elevation and subsequent restoration will be done using bioactive goimer material
  Interventions: Other: Assigned Interventions

INTERVENTIONS:
Other: Assigned Interventions — SDR Smart dentine replacement material nonbioactive

SUMMARY:
Deep marginal elevation usinge a bioactive dental material in deep subgingival Class II restorations, S-PRG filler-containing materials offer significant benefits due to their bioactive properties, Their ability to release fluoride, remineralization potential and acid neutralization, reducing the risk of recurrent caries, particularly at the gingival margin(Imazato et al. 2023). The antibacterial and antifungal effects help inhibit biofilm formation, enhancing the longevity of restorations. Additionally, these materials support better marginal adaptation by reducing microleakage and improving bond durability (Imazato et al. 2023) This type of composite may improve the outcomes of deep subgingival margin elevation, benefiting both restorative success and periodontal health(Imazato et al. 2023).

ELIGIBILITY:
Inclusion Criteria:

* Adults patients (20-50)
* Good oral hygiene (plaque index 0 or 1 )
* Patient approving to participate in the study
* Absence of parafunctional habits and/or bruxism
* No sign of irreversible pulpitis
* No periapical radiolucency
* Deep subgingival margin
* Molars class II with subgingival margin

Exclusion Criteria:

* • Patients with known allergic or adverse reaction to the tested materials.

  * Systematic disease that may affect participation.
  * Xerostomic patients.
  * Bad oral hygiene (plaque index 2 or 3 )
  * Heavy smokers
  * Patients undergoing or will start orthodontic treatment
  * Patients with removable prothesis

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-03-20 (Estimated); Primary Completion 2026-04-20 (Estimated); Study Completion 2026-04-20 (Estimated)

PRIMARY OUTCOMES:
Recurrent caries | T0: 1 Week Baseline T1: 6 Months T2: 12 Months
  * 0: no evidence of caries continuous along the margin using periapical radiograph.
  * 1: caries evident continuous with the margin of restoration

SECONDARY OUTCOMES:
Fracture of Restoration | T0: 1 Week Baseline T1: 6 Months T2: 12 Months
  * 1: Restoration is intact and fully retained.
  * 2:Restoration is partially retained with some portion of the restoration still intact.
  * 3:Restoration is completely missing
Post- operative sensitivity | T0: 1 Week Baseline T1: 6 Months T2: 12 Months
  * 1: Absent
  * 2: Present
Bleeding on Probing | T0: 1 Week Baseline T1: 6 Months T2: 12 Months
  * 0 :Healthy gums
  * 1 :Bleeding on probing

REFERENCES:
- [Background] Felemban MF, Khattak O, Alsharari T, Alzahrani AH, Ganji KK, Iqbal A. Relationship between Deep Marginal Elevation and Periodontal Parameters: A Systematic Review. Medicina (Kaunas). 2023 Nov 3;59(11):1948. doi: 10.3390/medicina59111948. PMID 38003997
- [Background] Choudhury WR, Nekkanti S. Mechanical Properties of SDR and Biodentine as Dentin Replacement Materials: An In Vitro Study. J Contemp Dent Pract. 2022 Jan 1;23(1):43-48. PMID 35656656